CLINICAL TRIAL: NCT07074093
Title: Effect of an Educational Intervention and an App-based Outdoor Air Pollution Alert System on Reducing Exacerbations in COPD Patients
Brief Title: Effect of an App-based Intervention on Air Pollution in COPD Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GRS 2519/B/22
Record Dates: First submitted 2025-07-08; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Air Quality; Mobile Health (mHealth); Digital Intervention; Smart Band / Wearable Device
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Intervention (Experimental): Participants will receive:
  COPD health education
  Training on and use of the AirVisual mobile app (real-time air quality info)
  Use of the Amazfit Band 5 (smart band to monitor activity and sleep)
  Usual COPD care
  Interventions: Combination Product: app+smartband+education
- Standard Care (No Intervention): Participants will receive:
  Usual COPD care and advice as per standard guidelines

INTERVENTIONS:
Combination Product: app+smartband+education — Intervention:
  Behavioral: Health education
  Device: AirVisual App
  Device: Amazfit Band 5
  Arms: Combined Intervention

SUMMARY:
This study will test whether a combination of health education, a mobile app, and a smart band can help people with chronic obstructive pulmonary disease (COPD) improve their quality of life and reduce flare-ups.

Participants will be randomly assigned to one of two groups:

One group will receive health education, use a mobile app that shows real-time air quality (AirVisual), and wear a smart band that tracks activity and sleep (Amazfit Band 5).

The other group will receive standard care and advice.

All participants will complete health checks and quality-of-life questionnaires at the beginning of the study and again after 6 months.

The goal is to find out if this combination of tools helps people with COPD manage their condition better and have fewer flare-ups.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a long-term lung condition that makes it hard to breathe and often gets worse over time. Many people with COPD experience flare-ups, which are periods when symptoms suddenly get worse. These flare-ups can be triggered by poor air quality and may lead to hospital visits or reduced quality of life.

This study will test a non-drug approach to help people with COPD manage their condition better. The researchers want to find out if using a combination of tools-health education, a mobile app, and a smart band-can reduce the number of flare-ups and improve quality of life.

The mobile app (AirVisual) provides real-time information about outdoor air quality, which may help participants avoid pollution. The smart band (Amazfit Band 5) tracks physical activity and sleep, helping users stay active and monitor their health. Participants in the intervention group will be trained on how to use both tools and receive general education about COPD management. The control group will receive standard care and advice.

A total of 150 participants will be recruited from urban health centers in Salamanca, Spain. Participants will be randomly assigned to either the intervention or control group. The study will last 6 months. All participants will have a clinical visit at the beginning and at the end of the study, where health measurements and quality-of-life questionnaires will be completed.

The goal is to learn whether this digital, non-pharmacological approach can support better daily management of COPD and lead to fewer symptom flare-ups.

ELIGIBILITY:
Inclusion Criteria:

Male or female, aged 18 years or older

Clinical diagnosis of chronic obstructive pulmonary disease (COPD) based on GOLD 2022 criteria (post-bronchodilator FEV1/FVC < 0.70)

Receiving care at urban primary care centers in Salamanca, Spain

Able to use a smartphone (independently or with minimal assistance)

Able and willing to provide written informed consent

Exclusion Criteria:

Diagnosis of a respiratory disease other than COPD (e.g., asthma, interstitial lung disease)

Moderate to severe cognitive impairment

Significant physical limitation that prevents participation in physical activity (e.g., NYHA Class III or IV heart failure, musculoskeletal conditions limiting walking)

Advanced kidney or liver disease

Severe mental illness or terminal condition

Participation in another clinical trial

Inability to use the mobile phone or smart band due to physical or technological limitations

Plans to relocate to another city within 12 months of study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of COPD exacerbations | From baseline to 6 months
  Number of moderate or severe exacerbations, defined as worsening of respiratory symptoms requiring systemic corticosteroids, antibiotics, or hospitalization.

SECONDARY OUTCOMES:
Change in health-related quality of life | Baseline and 6 months
  The Saint George's Respiratory Questionnaire assesses symptoms, activity limitation, and disease impact. Scores range from 0 (best health) to 100 (worst health).
Change in Physical Activity Level | Baseline to 6 months
  Global Physical Activity Questionnaire (GPAQ) in both groups; Step count and kilocalories burned (intervention group only, via Amazfit Band 5)
Change in BODE Index Score | Baseline and 6 months
  It stands for Body mass index, Obstruction (FEV1), Dyspnea (mMRC), and Exercise capacity (6-minute walk test). Its value ranges from 0 to 10 points, where 10 indicates maximum mortality risk. This score is divided into four quartiles to determine survival rates: quartile 1 (0-2 points - 82%), quartile 2 (3-4 points - 69%), quartile 3 (5-6 points - 60%), quartile 4 (7-10 points - 25%)
Change in Blood Pressure | Baseline and 6 months
  OMROM M10 blood pressure monitor (average of last 2 out of 3 measurements). SBP and DBP. Units: mmHg
Change in Lipid profile | Baseline and 6 months
  Total cholesterol, HDL, LDL, and triglycerides. Units: mg/dL
Healthcare Resource Use | 12 months before and 6 months after the intervention
  Number of primary care visits, emergency visits, hospital admissions, use of antibiotics, inhalers, and systemic corticosteroids (from Castilla y León EHR system)
Change in HbA1c | Baseline and 6 months
  A blood test that shows your average level of blood glucose over the past two to three months.

OTHER OUTCOMES:
Sex | Baseline
  Sex will be recorded as reported by the participant or as documented in the medical record. Categories: Male, Female
Body weight | Baseline and 6 months
  Measured with an electronic scale. Units: Kg
Height | Baseline and 6 months
  Measured using a calibrated stadiometer. Units: m
Frailty (for participants aged >65 years) | Baseline and 6 months
  Fried Frailty Criteria is a clinical scale used to assess frailty in older adults based on five components. Minimum and Maximum Values: 0-5. A higher score indicates greater frailty (0: Non-frail; 1-2: Pre-frail; 3-5: Frail)
ICT Usability and Adherence (Intervention Group only) | At 6 months
  mHealth App Usability Questionnaire (MAUQ) to assess the usability of the mobile health app. Contains multiple items rated on a 7-point Likert scale.
  Scores ranged from 20 to 140, and higher scores indicate better outcomes (greater usability and acceptance of the mobile app).
Smoking status | Baseline and 6 months
  Participants will be classified into three categories based on current and past smoking behaviour: Current smoker, Former smoker, Never smoker.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Investigación de AP de Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
PD Description: De-identified individual participant data that underlie the results reported in publications will be shared, including baseline characteristics, outcome measures, and limited subsets of laboratory and device-recorded data.
Supporting Information: Study Protocol
Time Frame: The protocol will be published by the end of 2025. De-identified participant data will be made available by the end of 2026, following the main results publication.
Access Criteria: Access will be granted to researchers whose proposed use of the data has been approved by an independent review committee identified for this purpose. Proposals should be directed to the corresponding author. Requestors will need to sign a data access agreement.
  Final access mechanism (repository or institutional platform) will be detailed upon publication.

REFERENCES:
- [Derived] Vicente-Garcia T, Maderuelo-Fernandez JA, Marcos-Romero I, Herrero-Hernandez B, Conde-Martin S, Rodriguez-Sanchez E, Gomez-Marcos MA, Garcia-Ortiz L, Lugones-Sanchez C. The effect of an educational intervention and an app-based outdoor air pollution alert system in reducing exacerbations in patients with COPD. BMC Prim Care. 2025 Dec 1;27(1):4. doi: 10.1186/s12875-025-03109-0. PMID 41327038